CLINICAL TRIAL: NCT00335985
Title: A Randomized, Double-blind, Controlled Clinical Study of GB-0998 for the Steroid-resistant Polymyositis and Dermatomyositis
Brief Title: Efficacy and Safety Study of GB-0998 for Treatment of Steroid-resistant Polymyositis and Dermatomyositis (PM/DM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Blood Products Organization (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0998-12
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2012-02

CONDITIONS: Polymyositis; Dermatomyositis
Keywords: polymyositis, dermatomyositis; High-dose intravenous immunoglobulin; Venoglobulin-IH; Steroid-resistant polymyositis(PM) and dermatomyositis(DM)
MeSH Terms: conditions — Polymyositis; Dermatomyositis | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: GB-0998
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo of GB-0998

INTERVENTIONS:
Drug: GB-0998 — 8 mL (400 mg of GB-0998)/kg per day is intravenously administered for five successive days
  Other Names: High-dose intravenous immunoglobulin; Venoglobulin-IH
  Arms: 1
Drug: Placebo of GB-0998 — 8 mL/kg per day is intravenously administered for five successive days
  Arms: 2

SUMMARY:
This randomized, double-blind, placebo-controlled trial will carry out to assess the efficacy of GB-0998 in the treatment of the steroid-resistant polymyositis and dermatomyositis based on the changes in manual muscle strength (MMT) scores as primary endpoint, and in addition, to assess the safety of GB-0998.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been defined as "definite" based on the criteria of Bohan and Peter for polymyositis and dermatomyositis.
* Patients who are defined as steroid-resistant ones based on the changes of scores on manual muscle testing (MMT) and serum levels of creatine kinase (CK) during observation period before administration of drug.

Exclusion Criteria:

* Patients with malignant tumors.
* Patients with acute interstitial pneumonia, including acute exacerbation of chronic.
* Patients with severe muscular atrophy for a long period.
* Patients with severe infectious disease.
* Patients who have the anamnesis of shock or hypersensitivity to this drug.
* Patients with severe hepatic disorder or severe renal disorder.
* Patients who have the anamnesis of cerebral infarction or ischemic heart disease, or who having symptom of these diseases.
* Patients who have been diagnosed as IgA deficiency in their past history.
* Pregnant, lactating, and probably pregnant patients, and patients who want to become pregnant.
* Patients who were administered immunoglobulin dosage within 6 weeks before consent.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Changes in manual muscle strength (MMT) scores | 8 weeks

SECONDARY OUTCOMES:
Changes in the serum levels of creatine kinase (CK) and total scores of activities of daily living (ADL) | 8 weeks
Adverse events and laboratory tests | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nobuyuki Miyasaka, Professor, Study Chair — Tokyo Medical and Dental University
Locations (1):
- Tokyo Medical and Dental University, Bunkyo-ku, Tokyo, Japan